CLINICAL TRIAL: NCT03846544
Title: Double Trigger and Ovum Retrieval vs. Conventional Antagonist Ovarian Stimulation Protocol in Poor Prognosis Women Undergoing IVF/ICSI: A Pilot Randomized Study
Brief Title: Double Pick up in Poor Prognosis Women
Acronym: DUOPICK
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: CRG UZ Brussel (Other)
Responsible Party: Principal Investigator, Panagiotis Drakopoulos, Prof. Dr., CRG UZ Brussel
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 58335
Record Dates: First submitted 2019-02-15; First posted 2019-02-19 (Actual); Results first posted 2024-04-15 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-04

CONDITIONS: Fertility Disorders

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (No Intervention)
- double pick up group (Experimental)
  Interventions: Drug: Corifollitoropin alfa (CFA)-double pick up

INTERVENTIONS:
Drug: Corifollitoropin alfa (CFA)-double pick up — In the study group, 225 IU of recombinant FSH (rFSH) will continue after the first oocyte retrieval (OR). Antagonist administration will be initiated when at least one follicle measuring ≥14 mm will be present in the ultrasound. If one or more follicles ≥17 mm are observed, patients will undergo a second triggering with human chorionic gonadotropin (hCG) 5000 IU and a second OR will be performed. In case of patients with no follicular development following 10 additional days of rFSH post-OR
  Arms: double pick up group

SUMMARY:
The purpose of this randomized pilot study is to compare the efficacy of double oocyte retrieval vs. conventional antagonist ovarian stimulation protocol in poor prognosis patients undergoing in vitro fertilization (IVF) or intra-cytoplasmic sperm injection (ICSI).

ELIGIBILITY:
Inclusion Criteria:

* Age 25-40 years
* Body mass index (BMI) ≤ 35 and ≥ 19
* Antimüllerian hormone (AMH) level of ≤1.5 ng/mL or antral follicular count (AFC) of ≤6 follicles or ≤5 oocytes retrieved in a previous cycle following standard conventional ovarian stimulation.

Exclusion Criteria:

* Testicular sperm extraction
* History of > 3 three consecutive previous unsuccessful IVF cycles
* BMI >35 or <19
* Use of oral contraceptives <3 months before start of the treatment
* polycystic ovary syndrome (PCOS) according to the Rotterdam criteria
* Ovarian stimulation for pre-implantation genetic testing (PGT-A/M)
* Medical/social freezing
* In vitro maturation (IVM)
* History of untreated autoimmune, endocrine or metabolic disorders,
* Ovarian cystectomy or oophorectomy

Ages: 25 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2021-09-15 (Actual); Study Completion 2022-10-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- UZ Brussel, Brussels, Jette, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Boudry L, Mateizel I, Wouters K, Papaleo E, Mackens S, De Vos M, Racca A, Adriaenssens T, Tournaye H, Blockeel C. Does dual oocyte retrieval with continuous FSH administration increase the number of mature oocytes in low responders? An open-label randomized controlled trial. Hum Reprod. 2024 Mar 1;39(3):538-547. doi: 10.1093/humrep/dead276. PMID 38199789

RESULTS

PARTICIPANT FLOW:
Groups:
- Control Group: conventional stimulation group
- Double Pick up Group: CFA-double pick up: In the study group, 225 IU of rFSH will continue after the first oocyte retrieval (OR). Antagonist administration will be initiated when at least one follicle measuring ≥14 mm will be present in the ultrasound. If one or more follicles ≥17 mm are observed, patients will undergo a second triggering with hCG 5000 IU and a second OR will be performed. In case of patients with no follicular development following 10 additional days of rFSH post-OR
Period: Overall Study
Arm/Group | Control Group | Double Pick up Group
Started | 24 | 24
Completed | 23 | 23
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Control Group: A single injection of 150mcg of corifollitropin alfa was administrated at day 2/3 of the cycle, followed by 225IU of recombinant FSH (rFSH) in a fixed antagonist protocol. Group A (control group) underwent conventional triggering with hCG 5000 IU and a single oocyte retrieval (OR)
- Double Pick up Group: A single injection of 150mcg of corifollitropin alfa was administrated at day 2/3 of the cycle, followed by 225IU of recombinant FSH (rFSH) in a fixed antagonist protocol. Group B (study group) underwent triggering with GnRHagonist. 225 IU of rFSH was continued after the first oocyte retrieval (OR). Antagonist administration was initiated when at least one follicle measuring ≥14 mm was present on the ultrasound. If one or more follicles ≥17 mm were observed, patients underwent a second triggering with hCG 5000 IU and a second OR was performed. In case of patients with no follicular development following 13 additional days of rFSH.
- Total: Total of all reporting groups
Arm/Group | Control Group | Double Pick up Group | Total
Number analyzed (Participants) | 24 | 24 | 48
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.3 (3.6) | 35.6 (2.9) | 36 (3.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 24 | 48
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 24 | 24 | 48
Body Mass index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 24.3 (3.7) | 24.5 (5.0) | 24.4 (4.3)
Anti-Müllerian hormone (AMH) [Mean (Standard Deviation); unit: ng/ml] | 0.5 (0.2) | 0.6 (0.3) | 0.55 (0.27)
antral follicle count (AFC) [Mean (Standard Deviation); unit: number of follicles] | 6.6 (3.3) | 5.7 (2.8) | 6.1 (3.1)
basal FSH [Mean (Standard Deviation); unit: IU/L] | 9.7 (3.6) | 9.8 (3.4) | 9.8 (3.4)
infertility duration [Mean (Standard Deviation); unit: years] | 2.4 (1.8) | 3.7 (7.0) | 3.1 (5.1)

OUTCOME MEASURES:

1. Primary Outcome: Number of MII Oocytes Retrieved Between the Two Arms
Description: number of mature (or metaphase II, MII) oocytes retrieved during oocyte retrieval
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: number of oocytes
Arm/Group | Control Group | Double Pick up Group
Number analyzed (Participants) | 23 | 23
number of oocytes | 4.1 (2.4) | 3.0 (2.2)

2. Secondary Outcome: Number of Preovulatory Follicles
Description: number of follicles ≥11m on the day of final oocyte maturation trigger
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: number of follicles
Arm/Group | Control Group | Double Pick up Group
Number analyzed (Participants) | 23 | 23
number of follicles | 5.4 (2.2) | 5.0 (1.6)

3. Secondary Outcome: Number of Cumulus Oocyte Complexes (COCs) Retrieved
Description: number of COCs retrieved at oocyte retrieval
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: number of oocytes
Arm/Group | Control Group | Double Pick up Group
Number analyzed (Participants) | 23 | 23
number of oocytes | 5.3 (2.7) | 3.3 (2.2)

4. Secondary Outcome: Number of Oocytes Fertilized
Description: number of fertilized oocytes at day 1 after oocyte retrieval
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: number of fertilized oocytes
Groups:
- Control Group: control group
Arm/Group | Control Group | Double Pick up Group
Number analyzed (Participants) | 23 | 23
number of fertilized oocytes | 3.7 (2.4) | 2.3 (2.0)

5. Secondary Outcome: Total Number of Available Embryos
Description: number of available embryos at day 3 or day 5 after oocyte retrieval, good quality and therefore transferable
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: number of embryos
Arm/Group | Control Group | Double Pick up Group
Number analyzed (Participants) | 23 | 23
number of embryos | 1.5 (0.9) | 1.4 (1.3)

6. Secondary Outcome: Duration of Ovarian Stimulation
Description: number of days of ovarian stimulation
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Control Group | Double Pick up Group
Number analyzed (Participants) | 23 | 23
days | 9.9 (2.7) | 9.9 (3.0)

7. Secondary Outcome: Clinical Pregnancy Rates
Description: clinical pregnancy rate
Time Frame: 4 months
Measure: Count of Participants; unit: Participants
Arm/Group | Control Group | Double Pick up Group
Number analyzed (Participants) | 23 | 23
Participants | 7 | 13

8. Secondary Outcome: Live Birth Rates
Description: number of live births
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Control Group | Double Pick up Group
Number analyzed (Participants) | 23 | 23
Participants | 6 | 8

9. Secondary Outcome: Cumulative Live Birth Rates
Description: defined as the first live birth following the transfer of fresh and subsequent frozen-thawed embryos
Time Frame: 24 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Control Group | Double Pick up Group
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/24
Other Adverse Events (participants affected / at risk) | 0/24 | 0/24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-06-03): https://cdn.clinicaltrials.gov/large-docs/44/NCT03846544/Prot_SAP_000.pdf